CLINICAL TRIAL: NCT05974618
Title: Prospective Validation of the ADNEX Model for Discrimination Between Benign and Malignant Adnexal Masses in Pregnancy: the International Ovarian Tumour Analysis in Pregnancy Study (p-IOTA).
Brief Title: Prospective Validation of the ADNEX Model for Discrimination Between Benign and Malignant Adnexal Masses in Pregnancy: International Ovarian Tumour Analysis in Pregnancy Study (p-IOTA)
Acronym: pIOTA
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S66455
Record Dates: First submitted 2023-07-10; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Adnexal Mass; Adnexal Tumor; Adnexal Cyst; Pregnancy Related
Keywords: IOTA; ovarian mass; pregnancy; ultrasound; post-partum; benign; malignant
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- First arm (primary objective):: First arm (primary objective): Adnexal mass scanned at 11-14 weeks. If the decision is to manage the adnexal mass conservatively, the patient is to be re-scanned once more: 0 - 90 days postpartum. In addition, the patient will be asked to enter into the third arm of the study (see below) knowing that she can opt out from that arm at any point. If she consents to participate in the third arm, she will participate in a series of longitudinal examinations as described for the third arm.
  All patients with a mass detected before 11 weeks will also be scanned at 11-14 weeks and can enter all three arms of the study. In this scenario, if more than one scan is performed during pregnancy before 11 weeks, only the first of several scans before 11 weeks will be included for the second and third arms of the study.
  Interventions: Diagnostic Test: Ultrasound
- Second arm (secondary objective):: Second arm (secondary objective): Adnexal mass is seen for the first time during that pregnancy at any gestation. If the decision is to manage the adnexal mass conservatively, the patient is to be re-scanned once more: 0 - 90 days postpartum. For patients with a mass detected before 11 weeks, see also above (they will be re-scanned at both 11-14 weeks and at 0-90 days postpartum).
  In addition, the patient will be asked to enter into the third arm of the study knowing that she can opt out from that arm at any point. If she consents to this, she will participate in a series of longitudinal examinations as described for the third arm.
  Interventions: Diagnostic Test: Ultrasound
- Third arm (secondary objective):: Third arm (secondary objective): Patients from the first and second arms who agree to enrol into the third arm i.e. longitudinal examination of an adnexal mass during pregnancy. For the purposes of the longitudinal evaluation, the time points for the ultrasound examination are:
  * initial presenting scan if <11 weeks;
  * 11-14 weeks;
  * 16 week scan - endometriomas ONLY;
  * second trimester routine scan (18-22 weeks);
  * 30-34 weeks;
  * any additional scans during pregnancy which resulted in either conservative management with extra scans or surgical intervention (with reason for the extra scan or for surgery documented);
  * 0-90 days postpartum.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — A standardised transvaginal (supplemented with transabdominal if transvaginal is not sufficient) examination is performed. When a colour Doppler ultrasound examination is performed, the pulse repetition frequency should be 0.3-0.6 KHz. The colour Doppler gain should be increased until colour Doppler artefacts appear and then lowered until just below the reappearance of colour Doppler artefacts. Ultrasound frequency and "priority" (grey scale or colour/Power Doppler) must also be optimised when using colour/power Doppler. Doppler ultrasound should be used with all masses included, irrespective of gestational age.

SUMMARY:
Prospective Validation of the ADNEX Model for discrimination between benign and malignant adnexal masses in pregnancy:

International Ovarian Tumour Analysis in pregnancy study (p-IOTA)

DETAILED DESCRIPTION:
1. STUDY SUMMARY

TITLE Prospective Validation of the ADNEX Model for discrimination between benign and malignant adnexal masses in pregnancy: the International Ovarian Tumour Analysis in pregnancy study (p-IOTA).

DESIGN Multicentre, prospective cohort observational study.

BACKGROUND Adnexal masses are a common incidental finding in pregnancy. Whilst the majority are benign and resolve spontaneously, a proportion can exhibit suspicious features during pregnancy raising concern about an underlying malignancy. Correct classification of adnexal masses is particularly important during pregnancy given the potential foetal and maternal risks associated with surgical intervention. International Ovarian Tumour Analysis (IOTA) group have developed robust, ultrasound-based tools, including the ADNEX model to support the classification of adnexal masses. Ultrasound-based tools such the Modified Benign Simple Descriptors and ADNEX have been externally validated to aid in the classification of adnexal masses in non-pregnant women, but their use as a robust diagnostic tool in pregnancy remains to be demonstrated.

AIMS The principal objective of this study is to prospectively investigate the ability of the ADNEX Model and a 2-step strategy (i.e. Modified Benign Simple Descriptors followed by ADNEX) to correctly discriminate between benign and malignant adnexal masses diagnosed in pregnancy.

PRIMARY OUTCOME MEASURE False discovery rate (number of benign masses / number of masses classified as malignant) when using the ADNEX Model to discriminate between benign and malignant adnexal masses at 11-14 gestational weeks in pregnancy.

ELIGIBILITY All women 18 years old and above with an adnexal mass found on ultrasound scan during pregnancy - irrespective of whether the mass known before pregnancy OR diagnosed for the first time on ultrasound scan during pregnancy.

DURATION This study will be conducted over a minimum period of three years.

KEYWORDS IOTA, ovarian mass, benign, malignant, ultrasound, pregnancy, post-partum

ELIGIBILITY:
Inclusion Criteria:

* • Consecutive patients with non-physiological adnexal masses or physiological cysts measuring 5cm or more in largest dimension;

  * In case of more than one mass seen, only most suspicious mass to be included OR in case of two similar masses, the one with the largest dimension or most easily accessible with ultrasound;
  * Previously recruited patient presenting with a different mass in subsequent pregnancy;
  * Age 18 years and above.

Exclusion Criteria:

* • Cysts deemed to be clearly physiological WHEN smaller than 5 cm (largest diameter);

  * Non-adnexal masses, e.g. peritoneal inclusion cysts (when diagnosis is certain) and peritoneal carcinomatosis with no adnexal mass;
  * The denial or withdrawal of written informed consent;
  * Same cyst already recruited for p-IOTA in a previous pregnancy.
  * Age < 18 years

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Our sample population will come from Early Pregnancy Units and from Tertiary referral centres for ultrasound with or without an oncology department attached to it. The sample size estimation is based on data from Tertiary referral centres.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
- Estimation of the false discovery rate when the ADNEX Model is applied at 11-14 weeks. | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  - Estimation of the false discovery rate when the ADNEX Model is applied at 11-14 weeks.

SECONDARY OUTCOMES:
- Estimation of the false discovery rate when the 2-step strategy (i.e. Modified Benign Simple Descriptors followed by ADNEX) is applied at 11-14 weeks. | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  - Estimation of the false discovery rate when the 2-step strategy (i.e. Modified Benign Simple Descriptors followed by ADNEX) is applied at 11-14 weeks.
- Estimation of the false discovery rate when the ADNEX Model and the 2-step strategy (i.e. Modified Benign Simple Descriptors followed by ADNEX) are applied at any time point during pregnancy; | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  - Estimation of the false discovery rate when the ADNEX Model and the 2-step strategy (i.e. Modified Benign Simple Descriptors followed by ADNEX) are applied at any time point during pregnancy;
Estimation of the ability of the ADNEX model and of the 2-step strategy to discriminate between benign and malignant adnexal masses when detected at 11-14 weeks gestation. | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  C-index
Estimation of the ability of the ADNEX model and of the 2-step strategy to discriminate between benign and malignant adnexal masses when detected at 11-14 weeks gestation. | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  (Sensitivity, Specificity)
Estimation of the ability of the ADNEX model and of the 2-step strategy to discriminate between benign and malignant adnexal masses when detected at 11-14 weeks gestation. | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  (Calibration)
Estimation of the ability of the ADNEX model and of the 2-step strategy to discriminate between benign and malignant adnexal masses when detected at 11-14 weeks gestation. | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  (Clinical utility) Net benefit.
Estimation of the ability of the ADNEX model and of the 2-step strategy to discriminate between benign and malignant adnexal masses when detected at any time point in pregnancy. | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  (C-index)
Estimation of the ability of the ADNEX model and of the 2-step strategy to discriminate between benign and malignant adnexal masses when detected at any time point in pregnancy. | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  (Sensitivity, Specificity)
Estimation of the ability of the ADNEX model and of the 2-step strategy to discriminate between benign and malignant adnexal masses when detected at any time point in pregnancy. | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  (Calibration)
Estimation of the ability of the ADNEX model and of the 2-step strategy to discriminate between benign and malignant adnexal masses when detected at any time point in pregnancy. | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  (Clinical utility) Net benefit.
- Estimation of the ability of the ADNEX model and the 2-step strategy to discriminate between benign and malignant adnexal masses when detected at any time po | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  - Estimation of the ability of the ADNEX model and the 2-step strategy (sensitivity, specificity, C-index, calibration intercept, calibration slope, clinical utility) to discriminate between benign and malignant adnexal masses when detected at any time point in pregnancy;
Evaluation of change in morphology of ovarian masses throughout pregnancy based on subjective assessment; | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  Evaluation of change in morphology of ovarian masses throughout pregnancy based on subjective assessment;
Evaluation of change throughout pregnancy and postpartum in papillations based on subjective assessment. | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  Number, size (mm), colour score (1-4), and morphology.

OTHER OUTCOMES:
Change in the ultrasound appearance of endometriomas during gestation; | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  Change in the ultrasound appearance of endometriomas during gestation;
- Occurrence of complications such as rupture, torsion, or malignancy during pregnancy in patients with conservatively treated masses (cumulative incidence illustrated by 'reverse' Kaplan-Meier curves). | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  - Occurrence of complications such as rupture, torsion, or malignancy during pregnancy in patients with conservatively treated masses (cumulative incidence illustrated by 'reverse' Kaplan-Meier curves).
- Comparison of the performance of ADNEX with CA125 and that of ADNEX without CA125. | outcome based on histology (surgery during pregnancy or within 120 days after postpartum ultrasound scan) or follow-up at postpartum scan (maximum one year after recruitment)
  (Specificity, Sensitivity, C-index, Calibration, Clinical Utility)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goh WA, Rincon M, Bohrer J, Tolosa JE, Sohaey R, Riano R, Davis J, Zalud I. Persistent ovarian masses and pregnancy outcomes. J Matern Fetal Neonatal Med. 2013 Jul;26(11):1090-3. doi: 10.3109/14767058.2013.768980. Epub 2013 Feb 21. PMID 23356452
- [Background] Sherard GB 3rd, Hodson CA, Williams HJ, Semer DA, Hadi HA, Tait DL. Adnexal masses and pregnancy: a 12-year experience. Am J Obstet Gynecol. 2003 Aug;189(2):358-62; discussion 362-3. doi: 10.1067/s0002-9378(03)00731-2. PMID 14520194
- [Background] Korenaga TK, Tewari KS. Gynecologic cancer in pregnancy. Gynecol Oncol. 2020 Jun;157(3):799-809. doi: 10.1016/j.ygyno.2020.03.015. Epub 2020 Apr 5. PMID 32268951
- [Background] de Haan J, Verheecke M, Van Calsteren K, Van Calster B, Shmakov RG, Mhallem Gziri M, Halaska MJ, Fruscio R, Lok CAR, Boere IA, Zola P, Ottevanger PB, de Groot CJM, Peccatori FA, Dahl Steffensen K, Cardonick EH, Polushkina E, Rob L, Ceppi L, Sukhikh GT, Han SN, Amant F; International Network on Cancer and Infertility Pregnancy (INCIP). Oncological management and obstetric and neonatal outcomes for women diagnosed with cancer during pregnancy: a 20-year international cohort study of 1170 patients. Lancet Oncol. 2018 Mar;19(3):337-346. doi: 10.1016/S1470-2045(18)30059-7. Epub 2018 Jan 26. PMID 29395867
- [Background] Leiserowitz GS, Xing G, Cress R, Brahmbhatt B, Dalrymple JL, Smith LH. Adnexal masses in pregnancy: how often are they malignant? Gynecol Oncol. 2006 May;101(2):315-21. doi: 10.1016/j.ygyno.2005.10.022. Epub 2005 Nov 28. PMID 16310839
- [Background] Froyman W, Landolfo C, De Cock B, Wynants L, Sladkevicius P, Testa AC, Van Holsbeke C, Domali E, Fruscio R, Epstein E, Dos Santos Bernardo MJ, Franchi D, Kudla MJ, Chiappa V, Alcazar JL, Leone FPG, Buonomo F, Hochberg L, Coccia ME, Guerriero S, Deo N, Jokubkiene L, Kaijser J, Coosemans A, Vergote I, Verbakel JY, Bourne T, Van Calster B, Valentin L, Timmerman D. Risk of complications in patients with conservatively managed ovarian tumours (IOTA5): a 2-year interim analysis of a multicentre, prospective, cohort study. Lancet Oncol. 2019 Mar;20(3):448-458. doi: 10.1016/S1470-2045(18)30837-4. Epub 2019 Feb 5. PMID 30737137
- [Background] Alcazar JL, Pascual MA, Graupera B, Auba M, Errasti T, Olartecoechea B, Ruiz-Zambrana A, Hereter L, Ajossa S, Guerriero S. External validation of IOTA simple descriptors and simple rules for classifying adnexal masses. Ultrasound Obstet Gynecol. 2016 Sep;48(3):397-402. doi: 10.1002/uog.15854. PMID 26748432
- [Background] Sayasneh A, Kaijser J, Preisler J, Johnson S, Stalder C, Husicka R, Guha S, Naji O, Abdallah Y, Raslan F, Drought A, Smith AA, Fotopoulou C, Ghaem-Maghami S, Van Calster B, Timmerman D, Bourne T. A multicenter prospective external validation of the diagnostic performance of IOTA simple descriptors and rules to characterize ovarian masses. Gynecol Oncol. 2013 Jul;130(1):140-6. doi: 10.1016/j.ygyno.2013.04.003. Epub 2013 Apr 8. PMID 23578539
- [Background] Sayasneh A, Ferrara L, De Cock B, Saso S, Al-Memar M, Johnson S, Kaijser J, Carvalho J, Husicka R, Smith A, Stalder C, Blanco MC, Ettore G, Van Calster B, Timmerman D, Bourne T. Evaluating the risk of ovarian cancer before surgery using the ADNEX model: a multicentre external validation study. Br J Cancer. 2016 Aug 23;115(5):542-8. doi: 10.1038/bjc.2016.227. Epub 2016 Aug 2. PMID 27482647
- [Background] Timmerman D, Testa AC, Bourne T, Ferrazzi E, Ameye L, Konstantinovic ML, Van Calster B, Collins WP, Vergote I, Van Huffel S, Valentin L; International Ovarian Tumor Analysis Group. Logistic regression model to distinguish between the benign and malignant adnexal mass before surgery: a multicenter study by the International Ovarian Tumor Analysis Group. J Clin Oncol. 2005 Dec 1;23(34):8794-801. doi: 10.1200/JCO.2005.01.7632. PMID 16314639
- [Background] Timmerman D, Van Calster B, Testa AC, Guerriero S, Fischerova D, Lissoni AA, Van Holsbeke C, Fruscio R, Czekierdowski A, Jurkovic D, Savelli L, Vergote I, Bourne T, Van Huffel S, Valentin L. Ovarian cancer prediction in adnexal masses using ultrasound-based logistic regression models: a temporal and external validation study by the IOTA group. Ultrasound Obstet Gynecol. 2010 Aug;36(2):226-34. doi: 10.1002/uog.7636. PMID 20455203
- [Background] Timmerman D, Ameye L, Fischerova D, Epstein E, Melis GB, Guerriero S, Van Holsbeke C, Savelli L, Fruscio R, Lissoni AA, Testa AC, Veldman J, Vergote I, Van Huffel S, Bourne T, Valentin L. Simple ultrasound rules to distinguish between benign and malignant adnexal masses before surgery: prospective validation by IOTA group. BMJ. 2010 Dec 14;341:c6839. doi: 10.1136/bmj.c6839. PMID 21156740
- [Background] Timmerman D, Van Calster B, Testa A, Savelli L, Fischerova D, Froyman W, Wynants L, Van Holsbeke C, Epstein E, Franchi D, Kaijser J, Czekierdowski A, Guerriero S, Fruscio R, Leone FPG, Rossi A, Landolfo C, Vergote I, Bourne T, Valentin L. Predicting the risk of malignancy in adnexal masses based on the Simple Rules from the International Ovarian Tumor Analysis group. Am J Obstet Gynecol. 2016 Apr;214(4):424-437. doi: 10.1016/j.ajog.2016.01.007. Epub 2016 Jan 19. PMID 26800772
- [Background] Van Calster B, Van Hoorde K, Valentin L, Testa AC, Fischerova D, Van Holsbeke C, Savelli L, Franchi D, Epstein E, Kaijser J, Van Belle V, Czekierdowski A, Guerriero S, Fruscio R, Lanzani C, Scala F, Bourne T, Timmerman D; International Ovarian Tumour Analysis Group. Evaluating the risk of ovarian cancer before surgery using the ADNEX model to differentiate between benign, borderline, early and advanced stage invasive, and secondary metastatic tumours: prospective multicentre diagnostic study. BMJ. 2014 Oct 15;349:g5920. doi: 10.1136/bmj.g5920. PMID 25320247
- [Background] Timmerman D, Testa AC, Bourne T, Ameye L, Jurkovic D, Van Holsbeke C, Paladini D, Van Calster B, Vergote I, Van Huffel S, Valentin L. Simple ultrasound-based rules for the diagnosis of ovarian cancer. Ultrasound Obstet Gynecol. 2008 Jun;31(6):681-90. doi: 10.1002/uog.5365. PMID 18504770
- [Background] Jacobs I, Oram D, Fairbanks J, Turner J, Frost C, Grudzinskas JG. A risk of malignancy index incorporating CA 125, ultrasound and menopausal status for the accurate preoperative diagnosis of ovarian cancer. Br J Obstet Gynaecol. 1990 Oct;97(10):922-9. doi: 10.1111/j.1471-0528.1990.tb02448.x. PMID 2223684
- [Background] Davies AP, Jacobs I, Woolas R, Fish A, Oram D. The adnexal mass: benign or malignant? Evaluation of a risk of malignancy index. Br J Obstet Gynaecol. 1993 Oct;100(10):927-31. doi: 10.1111/j.1471-0528.1993.tb15109.x. PMID 8217976
- [Background] Timmerman D, Van Calster B, Jurkovic D, Valentin L, Testa AC, Bernard JP, Van Holsbeke C, Van Huffel S, Vergote I, Bourne T. Inclusion of CA-125 does not improve mathematical models developed to distinguish between benign and malignant adnexal tumors. J Clin Oncol. 2007 Sep 20;25(27):4194-200. doi: 10.1200/JCO.2006.09.5943. Epub 2007 Aug 13. PMID 17698805
- [Background] Van Calster B, Timmerman D, Bourne T, Testa AC, Van Holsbeke C, Domali E, Jurkovic D, Neven P, Van Huffel S, Valentin L. Discrimination between benign and malignant adnexal masses by specialist ultrasound examination versus serum CA-125. J Natl Cancer Inst. 2007 Nov 21;99(22):1706-14. doi: 10.1093/jnci/djm199. Epub 2007 Nov 13. PMID 18000221
- [Background] Nustad K, Bast RC Jr, Brien TJ, Nilsson O, Seguin P, Suresh MR, Saga T, Nozawa S, Bormer OP, de Bruijn HW, Nap M, Vitali A, Gadnell M, Clark J, Shigemasa K, Karlsson B, Kreutz FT, Jette D, Sakahara H, Endo K, Paus E, Warren D, Hammarstrom S, Kenemans P, Hilgers J. Specificity and affinity of 26 monoclonal antibodies against the CA 125 antigen: first report from the ISOBM TD-1 workshop. International Society for Oncodevelopmental Biology and Medicine. Tumour Biol. 1996;17(4):196-219. doi: 10.1159/000217982. PMID 8685601
- [Background] Sarandakou A, Protonotariou E, Rizos D. Tumor markers in biological fluids associated with pregnancy. Crit Rev Clin Lab Sci. 2007;44(2):151-78. doi: 10.1080/10408360601003143. PMID 17364691
- [Background] Yazbek J, Salim R, Woelfer B, Aslam N, Lee CT, Jurkovic D. The value of ultrasound visualization of the ovaries during the routine 11-14 weeks nuchal translucency scan. Eur J Obstet Gynecol Reprod Biol. 2007 Jun;132(2):154-8. doi: 10.1016/j.ejogrb.2006.07.013. Epub 2006 Aug 17. PMID 16914254
- [Background] Mukhopadhyay A, Shinde A, Naik R. Ovarian cysts and cancer in pregnancy. Best Pract Res Clin Obstet Gynaecol. 2016 May;33:58-72. doi: 10.1016/j.bpobgyn.2015.10.015. Epub 2015 Oct 30. PMID 26707193
- [Background] Akazawa M, Onjo S. Malignant Transformation of Mature Cystic Teratoma: Is Squamous Cell Carcinoma Different From the Other Types of Neoplasm? Int J Gynecol Cancer. 2018 Nov;28(9):1650-1656. doi: 10.1097/IGC.0000000000001375. PMID 30358706
- [Background] Ayhan A, Aksu T, Develioglu O, Tuncer ZS, Ayhan A. Complications and bilaterality of mature ovarian teratomas (clinicopathological evaluation of 286 cases). Aust N Z J Obstet Gynaecol. 1991 Feb;31(1):83-5. doi: 10.1111/j.1479-828x.1991.tb02773.x. PMID 1872783
- [Background] Caspi B, Levi R, Appelman Z, Rabinerson D, Goldman G, Hagay Z. Conservative management of ovarian cystic teratoma during pregnancy and labor. Am J Obstet Gynecol. 2000 Mar;182(3):503-5. doi: 10.1067/mob.2000.103768. PMID 10739498
- [Background] Hoo WL, Yazbek J, Holland T, Mavrelos D, Tong EN, Jurkovic D. Expectant management of ultrasonically diagnosed ovarian dermoid cysts: is it possible to predict outcome? Ultrasound Obstet Gynecol. 2010 Aug;36(2):235-40. doi: 10.1002/uog.7610. PMID 20201114
- [Background] Caspi B, Appelman Z, Rabinerson D, Zalel Y, Tulandi T, Shoham Z. The growth pattern of ovarian dermoid cysts: a prospective study in premenopausal and postmenopausal women. Fertil Steril. 1997 Sep;68(3):501-5. doi: 10.1016/s0015-0282(97)00228-8. PMID 9314922
- [Background] Morice P. Borderline tumours of the ovary and fertility. Eur J Cancer. 2006 Jan;42(2):149-58. doi: 10.1016/j.ejca.2005.07.029. Epub 2005 Dec 2. PMID 16326097
- [Background] Hoover K, Jenkins TR. Evaluation and management of adnexal mass in pregnancy. Am J Obstet Gynecol. 2011 Aug;205(2):97-102. doi: 10.1016/j.ajog.2011.01.050. Epub 2011 May 14. PMID 21571247
- [Background] Fauvet R, Brzakowski M, Morice P, Resch B, Marret H, Graesslin O, Darai E. Borderline ovarian tumors diagnosed during pregnancy exhibit a high incidence of aggressive features: results of a French multicenter study. Ann Oncol. 2012 Jun;23(6):1481-7. doi: 10.1093/annonc/mdr452. Epub 2011 Oct 14. PMID 22003244
- [Background] Poder L, Coakley FV, Rabban JT, Goldstein RB, Aziz S, Chen LM. Decidualized endometrioma during pregnancy: recognizing an imaging mimic of ovarian malignancy. J Comput Assist Tomogr. 2008 Jul-Aug;32(4):555-8. doi: 10.1097/RCT.0b013e31814685ca. PMID 18664842
- [Background] Condous G, Khalid A, Okaro E, Bourne T. Should we be examining the ovaries in pregnancy? Prevalence and natural history of adnexal pathology detected at first-trimester sonography. Ultrasound Obstet Gynecol. 2004 Jul;24(1):62-6. doi: 10.1002/uog.1083. PMID 15229918
- [Background] Pateman K, Moro F, Mavrelos D, Foo X, Hoo WL, Jurkovic D. Natural history of ovarian endometrioma in pregnancy. BMC Womens Health. 2014 Oct 15;14:128. doi: 10.1186/1472-6874-14-128. PMID 25315259
- [Background] Mascilini F, Savelli L, Scifo MC, Exacoustos C, Timor-Tritsch IE, De Blasis I, Moruzzi MC, Pasciuto T, Scambia G, Valentin L, Testa AC. Ovarian masses with papillary projections diagnosed and removed during pregnancy: ultrasound features and histological diagnosis. Ultrasound Obstet Gynecol. 2017 Jul;50(1):116-123. doi: 10.1002/uog.17216. PMID 27484484
- [Background] Moro F, Mascilini F, Pasciuto T, Leombroni M, Li Destri M, De Blasis I, Garofalo S, Scambia G, Testa AC. Ultrasound features and clinical outcome of patients with malignant ovarian masses diagnosed during pregnancy: experience of a gynecological oncology ultrasound center. Int J Gynecol Cancer. 2019 Sep;29(7):1182-1194. doi: 10.1136/ijgc-2019-000373. Epub 2019 Jul 19. PMID 31326950
- [Background] Testa AC, Mascilini F, Quagliozzi L, Moro F, Bolomini G, Mirandola MT, Moruzzi MC, Scambia G, Fagotti A. Management of ovarian masses in pregnancy: patient selection for interventional treatment. Int J Gynecol Cancer. 2021 Jun;31(6):899-906. doi: 10.1136/ijgc-2020-001996. Epub 2020 Nov 10. PMID 33172924
- [Background] Hasson J, Tsafrir Z, Azem F, Bar-On S, Almog B, Mashiach R, Seidman D, Lessing JB, Grisaru D. Comparison of adnexal torsion between pregnant and nonpregnant women. Am J Obstet Gynecol. 2010 Jun;202(6):536.e1-6. doi: 10.1016/j.ajog.2009.11.028. Epub 2010 Jan 8. PMID 20060090
- [Background] Ginath S, Shalev A, Keidar R, Kerner R, Condrea A, Golan A, Sagiv R. Differences between adnexal torsion in pregnant and nonpregnant women. J Minim Invasive Gynecol. 2012 Nov-Dec;19(6):708-14. doi: 10.1016/j.jmig.2012.07.007. PMID 23084674
- [Background] Bignardi T, Condous G. The management of ovarian pathology in pregnancy. Best Pract Res Clin Obstet Gynaecol. 2009 Aug;23(4):539-48. doi: 10.1016/j.bpobgyn.2009.01.009. Epub 2009 Feb 20. PMID 19230784
- [Background] Yen CF, Lin SL, Murk W, Wang CJ, Lee CL, Soong YK, Arici A. Risk analysis of torsion and malignancy for adnexal masses during pregnancy. Fertil Steril. 2009 May;91(5):1895-902. doi: 10.1016/j.fertnstert.2008.02.014. Epub 2008 Mar 21. PMID 18359024
- [Background] Schmeler KM, Mayo-Smith WW, Peipert JF, Weitzen S, Manuel MD, Gordinier ME. Adnexal masses in pregnancy: surgery compared with observation. Obstet Gynecol. 2005 May;105(5 Pt 1):1098-103. doi: 10.1097/01.AOG.0000157465.99639.e5. PMID 15863550
- [Background] Germain A, Brunaud L. Visceral surgery and pregnancy. J Visc Surg. 2010 Jun;147(3):e129-35. doi: 10.1016/j.jviscsurg.2010.07.005. Epub 2010 Sep 1. PMID 20813621
- [Background] Balinskaite V, Bottle A, Sodhi V, Rivers A, Bennett PR, Brett SJ, Aylin P. The Risk of Adverse Pregnancy Outcomes Following Nonobstetric Surgery During Pregnancy: Estimates From a Retrospective Cohort Study of 6.5 Million Pregnancies. Ann Surg. 2017 Aug;266(2):260-266. doi: 10.1097/SLA.0000000000001976. PMID 27617856
- [Background] Soriano D, Yefet Y, Seidman DS, Goldenberg M, Mashiach S, Oelsner G. Laparoscopy versus laparotomy in the management of adnexal masses during pregnancy. Fertil Steril. 1999 May;71(5):955-60. doi: 10.1016/s0015-0282(99)00064-3. PMID 10231065
- [Background] Education and Practical Standards Committee, European Federation of Societies for Ultrasound in Medicine and Biology. Minimum training recommendations for the practice of medical ultrasound. Ultraschall Med. 2006 Feb;27(1):79-105. doi: 10.1055/s-2006-933605. No abstract available. PMID 16508866
- [Background] Riley RD, Debray TPA, Collins GS, Archer L, Ensor J, van Smeden M, Snell KIE. Minimum sample size for external validation of a clinical prediction model with a binary outcome. Stat Med. 2021 Aug 30;40(19):4230-4251. doi: 10.1002/sim.9025. Epub 2021 May 24. PMID 34031906

DOCUMENTS (2):
  • Study Protocol (2022-01-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT05974618/Prot_000.pdf
  • Informed Consent Form (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT05974618/ICF_001.pdf